CLINICAL TRIAL: NCT03790072
Title: Safety and Efficacy of Ex-vivo Expanded Allogeneic γδ T-lymphocytes (OmnImmune®) in Patients With Active Relapsed or Refractory Acute Myeloid Leukaemia (AML) Who Are Not Eligible for or do Not Consent to High Dose Salvage Chemotherapy and/or Allogeneic Haematopoietic Cell Transplantation (HCT). A Dose Escalation, Open-label, Phase I Study
Brief Title: Ex-vivo Expanded γδ T-lymphocytes (OmnImmune®) in Patients With Acute Myeloid Leukaemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TC Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TCB-202-001; 2018-000409-22 (EudraCT Number)
Record Dates: First submitted 2018-12-12; First posted 2018-12-31 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Gamma Delta T Lymphocytes
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Dose escalation, 3 cohorts, x10 dose increments between cohorts (10^6, 10^7, 10^8 of cells per kg of body weight).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): After inclusion, patients will receive conditioning chemotherapy consisting of non-investigational medicinal products (non-IMPs): fludarabine 25 mg/m2 from day -6 until day -2 (inclusive) and cyclophosphamide 500 mg/m2 on days -6 and -5.
  Subsequently, patients in will be dosed with investigational medicinal product (IMP) OmnImmune® on day 0.
  Interventions: Biological: OmnImmune®

INTERVENTIONS:
Biological: OmnImmune® — infusion of OmnImmune® (expanded gamma delta T lymphocytes)
  Other Names: fludarabine; cyclophosphamide

SUMMARY:
This study investigates the potential curative properties of gamma delta T-cells obtained from a blood-related donor of an AML patient.

DETAILED DESCRIPTION:
This is an open-label, safety and efficacy, escalating dose, single arm study on 9 adult subjects (3 cohorts) and 3+3 design will be used. HLA typed patients and potential blood-related donors will be screened for comorbidities. Suitably matched or haploidentical family donors will be selected according to protocol specified criteria and institutional guidelines of participating site.

ELIGIBILITY:
Inclusion Criteria:

1. History of acute myeloid leukaemia (initially diagnosed by presence of 20% or more blast cells with myeloid or monocytic differentiation confirmed by flow cytometry in peripheral blood or bone marrow)
2. Relapsed or refractory AML

   1. AML relapse after intensive chemotherapy OR
   2. AML relapse after allogeneic HCT OR
   3. AML progression on low intensity therapy (low dose cytarabine, 5-azacytidine or decitabine) OR
   4. No response to at least 4 cycles of low intensity therapy
   5. AML refractory to 2 cycles of induction chemotherapy
3. Presence of > 5% of blasts in bone marrow or peripheral blood smear
4. Patient not eligible for or does not consent to high dose salvage chemotherapy and/or allogeneic Haematopoietic Cell Transplantation (HCT)
5. Considered suitable for lymphodepleting chemotherapy
6. Age 18 years up to the age of 70 (≤ 70)
7. Life expectancy of at least 3 months
8. Karnofsky performance status ≥ 50%
9. Available related HLA-haploidentical or HLA-matched donor
10. Ability to be off systemic prednisone and other immunosuppressive drugs for at least 3 days prior to γδ T cells product infusion. Maintenance replacement steroid is allowed.
11. Patient able to understand and sign written informed consent

Exclusion Criteria:

1. Uncontrolled infections
2. Renal insufficiency: creatinine > 180 μmol/L or on dialysis
3. Heart failure: EF < 40%
4. Respiratory insufficiency: oxygen therapy required at inclusion in the study
5. Significant liver impairment: bilirubin > 50 μmol/L, AST or ALT > 4 times normal upper limit
6. Treatment with bisphosphonates (2 months before start)
7. Active autoimmune disease or GvHD
8. Pregnant or breastfeeding
9. Patient of fertile age not using two-barrier method of birth control.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AEs) [Safety] | Day 28 after completion of treatment
  Safety of OmnImmune® assessed by incidence of treatment-emergent adverse events (AEs) per patient graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Incidence of Dose-Limiting Toxicities (DLTs) [Tolerability] | Day 28 after completion of treatment
  Tolerability of OmnImmune® assessed by incidence of dose-limiting toxicities (DLTs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0

SECONDARY OUTCOMES:
Number of patients reaching Complete Remission (CR) [Efficacy] | 24 months post-treatment
  Efficacy of OmnImmune® assessed by number of patients reaching Complete Remission (CR)
Overall Survival (OS) [Efficacy] | 24 months post-treatment
  Efficacy of OmnImmune® assessed by overall survival (OS) measured in months
Quality of Life (QoL) | 24 months post-treatment
  Quality of life determined by European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire 'C30' which comprises 30 items (i.e. single questions), 24 of which are aggregated into nine multi-item scales, that is, five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

OTHER OUTCOMES:
Persistence of γδ T cells | Before treatment and up to 24 months after treatment
  Persistence of γδ T cells assessed by number and phenotype of γδ T cells using flow cytometry assay in peripheral blood and bone marrow from dosed patients
Phenotype of γδ T cells | Before treatment and up to 24 months after treatment
  Phenotype of γδ T cells assessed by flow cytometry assay in peripheral blood and bone marrow from dosed patients

CONTACTS AND LOCATIONS:
Locations (1):
- UHKT (Ustav hematologie a krevni transfuze), Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided